CLINICAL TRIAL: NCT06469151
Title: A Phase I Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of AZD5148 in Healthy Adults
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of AZD5148 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: D8820C00002
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants
Keywords: Pharmacokinetics; Clostridioides difficile infection (CDI); Placebo-controlled; Anti-drug antibodies (ADA)
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1: AZD5148 (dose 1) IM (Experimental): Participants will receive AZD5148 (dose 1) or matching placebo as an IM injection
  Interventions: Drug: AZD5148; Drug: Placebo
- Cohort 2a: AZD5148 (dose 2) IM (Experimental): Participants will receive AZD5148 (dose 2) or matching placebo as an IM injection
  Interventions: Drug: AZD5148; Drug: Placebo
- Cohort 2b: AZD5148 (dose 2) IM (Experimental): Participants of Chinese descent will receive AZD5148 (dose 2) or matching placebo as an IM injection
  Interventions: Drug: AZD5148; Drug: Placebo
- Cohort 3: AZD5148 (dose 2) IV (Experimental): Participants will receive AZD5148 (dose 2) or matching placebo as an IV bolus
  Interventions: Drug: AZD5148; Drug: Placebo
- Cohort 4a: AZD5148 (dose 3) IV (Experimental): Participants will receive AZD5148 (dose 3) or matching placebo as an IV bolus
  Interventions: Drug: AZD5148; Drug: Placebo
- Cohort 4b: AZD5148 (dose 3) IV (Experimental): Participants of Chinese descent will receive AZD5148 (dose 3) or matching placebo as an IV bolus
  Interventions: Drug: AZD5148; Drug: Placebo
- Cohort 5: AZD5148 (dose 4) IV (Experimental): Participants will receive AZD5148 (dose 4) or matching placebo as an IV bolus
  Interventions: Drug: AZD5148; Drug: Placebo

INTERVENTIONS:
Drug: AZD5148 — Participants will receive AZD5148 (dose 1, dose 2, dose 3 or dose 4) as an IM injection or IV bolus
Drug: Placebo — Participants will receive matching doses of placebo as an IM injection or IV bolus

SUMMARY:
The purpose of this study is to measure safety, tolerability, and pharmacokinetics (PK) of a single dose of AZD5148 administered via intravenous (IV) bolus or intramuscular (IM) injection in healthy participants

DETAILED DESCRIPTION:
This is a first in human study which will be conducted at four clinical units. Participants will be randomized to receive AZD5148, or placebo administered by intramuscular (IM) injection into the lateral thigh muscle or intravenous (IV) bolus (single, discrete dose of a drug).

This study will include 7 dose cohorts, two of which will include exclusively participants of Chinese descent, Cohort 2b and 4b. Each dose cohort will begin with a Sentinel Group of 2 participants randomized 1:1 (AZD5148:placebo). The participants in the Sentinel Group will undergo a safety monitoring period of 24 hours before the remaining participants in that cohort are dosed. If there would be no safety concerns, the remaining participants in the cohort will be dosed in a 9:1 ratio (AZD5148: placebo). Each participant will be involved in the study for up to 56 weeks (including Screening Period)

The study will comprise:

* A Screening Period of maximum 28 days (Day -28 to Day -1 inclusive).
* A Treatment and Follow-up Period lasting 12 months after the administration of the study drug.

  * Participants will be resident at the Clinical Unit from the day before study drug administration (Day -1) until all assessments are completed on Day 2.
  * A final Follow-up Visit will occur within 361 ± 14 days after the study drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants with suitable veins for cannulation or repeated venipuncture at the time of consent.
* All women must have a negative serum pregnancy test at the Screening Visit.
* Women of childbearing potential must have a negative urine pregnancy test on admission to the Clinical Unit.
* Women of childbearing potential must not be lactating and if heterosexually active must agree to use an approved method of highly effective contraception, to avoid pregnancy from 3 months prior to administration of the study drug and until 360 days after the dose of the study drug.
* Women of non-childbearing potential must be confirmed at the Screening Visit by fulfilling one of the following criteria:

  1. Postmenopausal defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments and follicular stimulating hormone (FSH) levels in the postmenopausal range.
  2. Documentation of irreversible surgical sterilization by complete hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation or tubal occlusion.
* Have a Body mass index ≥ 18.0 to ≤ 32.0 kg/m2 and weigh ≥ 45 kg and ≤ 110 kg.
* Willing and able to complete the Follow-up Period through Day 361.
* Healthy Chinese participants - participants of Chinese descent are eligible based on meeting all of the following specific criteria for these two cohorts (Cohorts 2b and 4b):

  1. Participant with Chinese ancestry, born in mainland China, Hong Kong, or Taiwan.
  2. Participant is the descendant of 4 ethnic Chinese grandparents and 2 ethnic Chinese parents.
  3. Participant has lived outside China for ≤ 10 years at the time of Screening.
  4. Exhibits no significant change in lifestyle, including diet, since leaving China.

Exclusion Criteria:

* History of any clinically important disease or disorder which may either put the participant at risk because of participation in the study or influence the results or the participant's ability to participate in the study.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study drug.
* History of malignancy other than treated non-melanoma skin cancers or locally treated cervical cancer in previous 5 years.
* Any medical history of symptomatic CDI within the prior 2 years.
* Any clinically important abnormalities in laboratory values, vital signs, clinical chemistry, hematology, or urinalysis results.
* Any positive result on Screening for serum Hepatitis B surface antigen (HBsAg) or Hepatitis C virus (HCV).
* Primary or acquired immunodeficiency, including HIV infection or due to drugs, including any course of glucocorticoid therapy exceeding 2 weeks of prednisone or equivalent within 6 months prior to Screening. Human immunodeficiency virus (HIV) testing must be negative at Screening Visit.
* Any clinically important abnormalities in rhythm, conduction, or morphology of the resting 12-lead electrocardiogram, at Screening.
* Known or suspected history of alcohol or drug abuse within the past 2 years that might affect assessments of safety or ability of participant to comply with all study requirements.
* Positive screen for drugs of abuse, or alcohol at Screening or Day -1.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity to drugs with a similar chemical structure or class to the study drug.
* History of previous hypersensitivity, infusion-related reaction, or severe adverse reaction following administration of monoclonal antibodies (mAbs).
* Previous receipt of a mAb within 6 months, or 5 antibody half-lives (whichever is longer), prior to the start of the study.
* Plasma donation within one month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months prior to the Screening Visit.
* Receipt of immunoglobulin or blood products, or expected receipt, within 6 months prior to Screening or expected to receive during the study.
* Clinically significant bleeding disorder (e.g., factor VIII deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture.
* Vulnerable participants, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs). | From Day -1 to Day 91
  To evaluate the safety and tolerability of AZD5148 administered as a single IV or IM dose to healthy adult participants.
Number of participants with serious adverse events (SAEs) and adverse events of special interest (AESIs) | From Screening (Day -28 to Day -1) to final Follow-up Visit (Day 361 ± 14)
  To evaluate the safety and tolerability of AZD5148 administered as a single IV or IM dose to healthy adult participants.

SECONDARY OUTCOMES:
Maximum observed drug concentration (Cmax) | From Day 1 until last Follow up visit (Day 361 ± 14 days)
  To evaluate the single dose PK of AZD5148.
Time to reach maximum observed concentration (tmax) | From Day 1 until last Follow up visit (Day 361 ± 14 days)
  To evaluate the single dose PK of AZD5148.
Time of last quantifiable concentration (tlast) | From Day 1 until last Follow up visit (Day 361 ± 14 days)
  To evaluate the single dose PK of AZD5148.
Terminal elimination half-life, estimated as (ln2)/λz (t1/2λz) | From Day 1 until last Follow up visit (Day 361 ± 14 days)
  To evaluate the single dose PK of AZD5148.
Area under concentration-curve from time 0 to the time of last quantifiable concentration (AUClast) | From Day 1 until last Follow up visit (Day 361 ± 14 days)
  To evaluate the single dose PK of AZD5148.
Area under concentration-time curve from time 0 extrapolated to infinity (AUCinf) | From Day 1 until last Follow up visit (Day 361 ± 14 days)
  To evaluate the single dose PK of AZD5148.
Volume of distribution at steady state (IV administration only) (Vss) | From Day 1 until last Follow up visit (Day 361 ± 14 days)
  To evaluate the single dose PK of AZD5148.
Volume of distribution at terminal phase (IV administration only) (Vz) | From Day 1 until last Follow up visit (Day 361 ± 14 days)
  To evaluate the single dose PK of AZD5148.
Systematic clearance (IV administration only) (CL) | From Day 1 until last Follow up visit (Day 361 ± 14 days)
  To evaluate the single dose PK of AZD5148.
Apparent total body clearance (IM administration only) (CL/F) | From Day 1 until last Follow up visit (Day 361 ± 14 days)
  To evaluate the single dose PK of AZD5148.
Apparent volume of distribution based on the terminal phase (IM administration only) (Vz/F) | From Day 1 until last Follow up visit (Day 361 ± 14 days)
  To evaluate the single dose PK of AZD5148.
Bioavailability for extravascular administration (IM administration only) (F) | From Day 1 until last Follow up visit (Day 361 ± 14 days)
  To evaluate the single dose PK of AZD5148.
Incidence of positive ADAs against AZD5148 in serum | Day 1 (pre-dose), Day 29, Day 91, Day 181 and Day 361
  To evaluate the ADA responses to a single IV or IM dose of AZD5148.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Research Site, Anniston, Alabama
  - Research Site, Glendale, California
  - Research Site, Baltimore, Maryland
  - Research Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/